CLINICAL TRIAL: NCT01377246
Title: A PROSPECTIVE, RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED CLINICAL TRIAL TO ASSESS THE EFFECTS OF LONG-ACTING SOMATOSTATIN (OCTREOTIDE LAR) THERAPY ON DISEASE PROGRESSION IN PATIENTS WITH AUTOSOMAL DOMINANT POLYCYSTIC KIDNEY DISEASE AND MODERATE TO SEVERE RENAL INSUFFICIENCY
Brief Title: Somatostatin In Patients With Autosomal Dominant Polycystic Kidney Disease And Moderate To Severe Renal Insufficiency
Acronym: ALADIN2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALADIN2; 2011-000138-12 (EudraCT Number)
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Somatostatin.; Polycystic kidney disease.; Renal insufficiency.
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Renal Insufficiency | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline solution. (Placebo Comparator)
  Interventions: Other: Saline solution.
- Octrotide-LAR (Experimental)
  Interventions: Drug: Octreotide-LAR

INTERVENTIONS:
Drug: Octreotide-LAR — 40 mg every 28 days (in two intragluteal 20 mg injections) for three years
  Arms: Octrotide-LAR
Other: Saline solution. — At the same volume of study drug every 28 days (in two intragluteal injections) for three years.
  Arms: Saline solution.

SUMMARY:
The general aim of the trial is to assess the efficacy of one year treatment with long-acting somatostatin analogue (Octreotide LAR) compared with placebo in slowing kidney and liver growth rate in patients with ADPKD and moderate/severe renal insufficiency and to assess whether and to which extent this translates into slower renal function decline over 3-year follow-up.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD), the most common hereditary cystic renal disease, has an incidence of 1 in 800 live births and account for 7-10% of patients on dialysis in developed countries. Clinically, ADPKD is characterized by renal and extra renal manifestations. In the kidneys, multiple cysts grow from distal and collecting tubular epithelial cells producing progressive renal enlargement with relatively initial stable renal functions. Thereafter, both tubular and secondary interstitial damage lead to faster renal loss and end-stage renal disease (ESRD) in approximately half of all patients affected in their fifth or sixth decade of life. More than 50% of the patients display hepatic cysts derived from cholangiocyte proliferation and fluid secretion. Pancreatic and intestinal cysts as well as increased risk of aortic aneurysms, heart-valve defects and sudden death due to rupture of intracerebral aneurysms are extra-renal manifestations.

Patients with ADPKD, at similar levels of proteinuria and blood pressure control, do not seem to benefit to the same extent of ACE inhibitor therapy and have faster decline in glomerular filtration rate (GFR) compared with other chronic kidney diseases. Thus, in ADPKD renoprotective interventions - in addition to achieving maximal reduction of arterial blood pressure and proteinuria, and limiting the effects of other potential disease progression promoters (such as dyslipidemia, chronic hyperglycemia, or smoking)- should also be specifically aimed to correct the dysregulation of epithelial cell growth, fluid secretion, and extracellular matrix deposition that is characteristic of this disease. Up to now, no specific therapies for ADPKD are available, but drugs like somatostatin, rapamycin, and tolvaptan targeting to growth and chloride secretion pathways are now being testing worldwide in some clinical trials.

We have performed some years ago a pilot prospective cross-over controlled study with long-acting somatostatin analog in patients with ADPKD and different degree of renal dysfunction. We found that in these patients, 6 month treatment with octreotide was safe, well tolerated, and slowed the time-dependent increase in total kidney volume to a significant extent compared to placebo. The net effect in kidney volume resulted from an action of the drug on cyst volume and on parenchyma volume. Moreover, more recent post-hoc analysis of the concomitant liver disease progression in the same ADPKD patients demonstrated a significant reduction in the total liver volume during octreotide treatment, not appreciably observed during placebo. Moreover, in the untreated ADPKD patients enrolled in our study, computed tomography evaluation of disease progression showed that the ratio of faintly contrast-enhanced parenchyma volume over total parenchyma volume strongly correlated with basal GFR and GFR changes during the observation period.

The good safety profile of octreotide and the slowing of renal growth demonstrated in our short-term clinical study did suggest the feasibility of a randomized trial in larger series of ADPKD patients with normal renal function or mild renal insufficiency to verify whether long-term somatostatin treatment may eventually provide effective renoprotection. This trial - the ALADIN study - is ongoing and the planned ADPKD patients have been enrolled. So far, no particular side effects have been reported. More important, preliminary interim analysis of data from patients who reached 1 year treatment, confirmed the beneficial effect of octreotide in slowing the growth of total kidney volume compared to placebo.

The findings of the safety and potential benefit of octreotide in few patients with severe renal insufficiency observed in our initial pilot study and the encouraging preliminary long-term effect results of octreotide on kidney growth, make worth investigating the efficacy of a long-acting somatostatin (Octreotide LAR) in slowing or even halting the kidney enlargement and renal function decline in ADPKD patients with moderate/severe renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical and ultrasound diagnosis of ADPKD
* Estimated GFR between 15 and 40 ml/min/1.73m2 (by the MDRD 4 variable equation)
* Written informed consent

Exclusion Criteria:

* 24-h Urinary protein excretion rate >3g (suggestive of a concomitant glomerular disease that could benefit of specific therapy)
* Symptomatic urinary tract lithiasis or obstruction
* Uncontrolled diabetes mellitus (HbA1c >8%) or hypertension (systolic/diastolic BP >180/110 mmHg)
* Current urinary tract infection
* Symptomatic biliary tract lithiasis
* Active cancer
* Psychiatric disorders or any condition that might prevent full comprehension of the purposes and risks of the study
* Pregnancy, lactation or child bearing potential and ineffective contraception (estrogen therapy in post menopausal women should not be stopped)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Total kidney volume (TKV) change (delta TKV) as assessed by spiral computed tomography (spiral CT) scan. | At 0, 12 and 36 month.
  Short-term (1 year)outcome.
Rate of GFR decline as assessed by serial measurements of the iohexol plasma clearance. | At 0, 12, 24 and 36 month.
  Long-term (3 year)outcome.

SECONDARY OUTCOMES:
Total renal cyst volume. | At 0,12 and 36 month.
Total renal parenchyma volume. | At 0, 12 and 36 month.
Total renal intermediate volume. | At 0,12 and 36 month.
Total liver and liver cyst volumes. | At 0, 12 and 36 month.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Ospedale San giovanni di Dio, Agrigento, AG
  - Clinical Research Center fo Rare Diseases Aldo and Cele Daccò, Ranica, Bergamo
  - Hospital "Vito Fazzi", Lecce
  - Hospital "Ospedale Maggiore policlinico, Mangiagalli e Regina elena", Milan
  - University "Federico II", Naples
  - Ospedale Cà Foncello, Treviso

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Perico N, Ruggenenti P, Perna A, Caroli A, Trillini M, Sironi S, Pisani A, Riccio E, Imbriaco M, Dugo M, Morana G, Granata A, Figuera M, Gaspari F, Carrara F, Rubis N, Villa A, Gamba S, Prandini S, Cortinovis M, Remuzzi A, Remuzzi G; ALADIN 2 Study Group. Octreotide-LAR in later-stage autosomal dominant polycystic kidney disease (ALADIN 2): A randomized, double-blind, placebo-controlled, multicenter trial. PLoS Med. 2019 Apr 5;16(4):e1002777. doi: 10.1371/journal.pmed.1002777. eCollection 2019 Apr. PMID 30951521